CLINICAL TRIAL: NCT04775472
Title: Early Left Atrial Septostomy Versus Conventional Approach After Venoarterial Extracorporeal Membrane Oxygenation: A Randomized Controlled Study
Brief Title: Early Left Atrial Septostomy Versus Conventional Approach After Venoarterial Extracorporeal Membrane Oxygenation
Acronym: EARLY-UNLOAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2020-390
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cardiogenic Shock
Keywords: Extracorporeal membrane oxygenation; Myocardial Infarction; Heart Diseases; Cardiovascular Diseases; Coronary Disease
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction; Heart Diseases; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early left atrial septostomy group (Experimental): Early left atrial septostomy group will routinely receive left atrial septostomy within 12 hours after VA-ECMO implantation.
  Interventions: Procedure: Early left atrial septostomy within 12 hours after VA-ECMO implantation
- Conventional approach group (Active Comparator): Conventional approach group will receive left atrial septostomy in cases of deleterious effect of increased LVEDP after VA-ECMO implantation, such as refractory pulmonary edema, abnormal opening of aortic valve, left ventricular dilatation, refractory ventricular tachycardia or fibrillation.
  Interventions: Procedure: Selective left atrial septostomy

INTERVENTIONS:
Procedure: Early left atrial septostomy within 12 hours after VA-ECMO implantation — Early left atrial septostomy group will routinely receive left atrial septostomy within 12 hours after VA-ECMO implantation. Left atrial septostomy will be done using percutaneous technique.
  Arms: Early left atrial septostomy group
Procedure: Selective left atrial septostomy — Left atrial septostomy will be done in cases of deleterious effect of increased LVEDP after VA-ECMO implantation, such as refractory pulmonary edema, abnormal opening of aortic valve, left ventricular dilatation, refractory ventricular tachycardia or fibrillation.
  Arms: Conventional approach group

SUMMARY:
The use of venoarterial-extracorporeal membrane oxygenation(VA-ECMO) was associated with lower in-hospital mortality in patients with cardiogenic shock. However, VA-ECMO has a deleterious effect for hemodynamics. It can increase left ventricular end-diastolic pressure(LVEDP), followed by left ventricular dilatation, abnormal opening of aortic valve and jeopardizes of myocardial recovery. Therefore, several methods have been used to reduce LVEDP. Among these, left atrial septostomy is effective, but less invasive than surgical left ventricular unloading. However, there is few data regarding this issue. Therefore, the investigators will evaluate the effect of routine, early left atrial septostomy in patients with VA-ECMO for the treatment of cardiogenic shock.

DETAILED DESCRIPTION:
Study Objectives:

To determine the effect of early left atrial septostomy versus conventional approach(left atrial septostomy only in cases of significant changes due to left ventricular end-diastolic pressure increase) in patients who received venoarterial-extracorporeal membrane oxygenation(VA-ECMO) for the treatment of cardiogenic shock.

Study Background:

Cardiogenic shock is due to myocardial dysfunction from multifactorial causes, which has high mortality. The treatment for cardiogenic shock includes early coronary revascularization, inotropes, vasopressors, or mechanical circulatory support, such as intraaortic balloon pump(IABP), VA-ECMO. However, the routine use of IABP is not recommended for the treatment of cardiogenic shock in recent guidelines. VA-ECMO can be easily implanted, and can maintain high cardiac output. In several studies, The use of VA-ECMO was associated with lower in-hospital mortality in patients with cardiogenic shock.

However, VA-ECMO has a deleterious effect for hemodynamics. It can increase left ventricular end-diastolic pressure(LVEDP), followed by left ventricular dilatation, abnormal opening of aortic valve and jeopardizes of myocardial recovery. Therefore, several methods have been used to reduce LVEDP. Among these, left atrial septostomy is effective, but less invasive than surgical left ventricular unloading. However, there is few data regarding this issue. Therefore, the investigators will evaluate the effect of routine, early left atrial septostomy in patients with VA-ECMO for the treatment of cardiogenic shock.

Study Hypothesis:

Early, routine left atrial septostomy for left heart unloading is superior compared to conventional approach to reduce in-hospital mortality and the duration of VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

1) Age more than 18 years old 2) Cardiogenic shock* 3) Successful VA-ECMO implantation

* The definition of cardiogenic shock All these criteria should be met

  1. Systolic blood pressure < 90 mmHg for 30 minutes, or needing inotrope or vasopressor to maintain systolic blood pressure > or = 90 mmHg
  2. Pulmonary congestion on chest X-ray or increased left ventricular filling pressure by cardiac catheterization
  3. At least one criteria of organ dysfunction

     - mental obtundation, clammy skin, oliguria, renal dysfunction, increased level of blood lactate

     Exclusion Criteria:

  <!-- -->

  1. VA-ECMO after open heart surgery
  2. VA-ECMO for the treatment of non-cardiac shock
  3. Severe bleeding*
  4. Terminal malignancy
  5. Irreversible brain damage
  6. Pregnancy or lactation
* The definition of severe bleeding Hemoglobin decrease after VA-ECMO or cannulation site bleeding is not a exclusion criteria

  1. Hypovolemic shock due to definite bleeding cause
  2. Identifiable bleeding causes: gastrointestinal bleeding, hemothorax, traumatic bleeding, central nervous system hemorrhage, pulmonary hemorrhage

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence rate of all-cause death | Up to 30 days
  Cumulative incidence rate of all-cause death

SECONDARY OUTCOMES:
Rate of all-cause death or left atrial septostomy in conventional approach group | Up to 30 days
  Rate of all-cause death or left atrial septostomy in conventional approach group
Rate of left atrial septostomy in conventional approach group | Up to 30 days
  Rate of left atrial septostomy in conventional approach group
Incidence rate of all-cause death during index admission | Up to 6 months
  Incidence rate of all-cause death during index admission
Cumulative incidence rate of cardiac death | Up to 30 days
  Cumulative incidence rate of cardiac death
Cumulative incidence rate of non-cardiac death | Up to 30 days
  Cumulative incidence rate of non-cardiac death
Weaning rate from venoarterial extracorporeal membrane oxygenation during index admission | Up to 6 months
  Weaning rate from venoarterial extracorporeal membrane oxygenation during index admission
Rate of disappearance of pulmonary edema on chest X-ray during index admission | Up to 6 months
  Rate of disappearance of pulmonary edema on chest X-ray during index admission
Weaning rate from mechanical ventilator during index admission | Up to 6 months
  Weaning rate from mechanical ventilator during index admission
Intensive care unit length of stay during index admission | Up to 6 months
  Intensive care unit length of stay during index admission
Hospital length of stay | Up to 6 months
  Hospital length of stay
Lactate normalization rate | Up to 30 days
  Lactate normalization rate
Lactate clearance rate | Up to 30 days
  Lactate clearance rate
Rate of renal replacement therapy during index admission | Up to 6 months
  Rate of renal replacement therapy during index admission
Rate of limb ischemia during index admission | Up to 6 months
  Rate of limb ischemia during index admission
Rate of infection during index admission | Up to 6 months
  Rate of infection during index admission
Rate of transient ischemic attack or stroke during index admission | Up to 6 months
  Rate of transient ischemic attack or stroke during index admission
Rate of BARC bleeding type 3 or 5 during index admission | Up to 6 months
  Rate of BARC bleeding type 3 or 5 during index admission
Rate of bridge to ventricular assist device or heart transplantation during index admission | Up to 6 months
  Rate of bridge to ventricular assist device or heart transplantation during index admission
Rate of major vascular injury or cardiac tamponade during left atrial septostomy | Up to 30 days
  Rate of major vascular injury or cardiac tamponade during left atrial septostomy
Cumulative incidence rate of all-cause death | Up to 12 months
  Cumulative incidence rate of all-cause death
Cumulative incidence rate of cardiac death | Up to 12 months
  Cumulative incidence rate of cardiac death
Cumulative incidence rate of non-cardiac death | Up to 12 months
  Cumulative incidence rate of non-cardiac death
Re-hospitalization rate due to heart failure | Up to 12 months
  Re-hospitalization rate due to heart failure
All-cause death or re-hospitalization rate due to heart failure | Up to 12 months
  All-cause death or re-hospitalization rate due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Kim, Professor, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim Y, Kim MC, Lee SH, Park S, Ahn JH, Hyun DY, Cho KH, Jung YH, Jeong IS, Ahn Y. Early left ventricular unloading after venoarterial extracorporeal membrane oxygenation: 1-year outcomes of the EARLY-UNLOAD randomized clinical trial. Eur Heart J Acute Cardiovasc Care. 2025 Apr 26;14(4):203-211. doi: 10.1093/ehjacc/zuae150. PMID 39749912
- [Derived] Kim MC, Lim Y, Lee SH, Shin Y, Ahn JH, Hyun DY, Cho KH, Sim DS, Hong YJ, Kim JH, Jeong MH, Jung YH, Jeong IS, Ahn Y. Early Left Ventricular Unloading or Conventional Approach After Venoarterial Extracorporeal Membrane Oxygenation: The EARLY-UNLOAD Randomized Clinical Trial. Circulation. 2023 Nov 14;148(20):1570-1581. doi: 10.1161/CIRCULATIONAHA.123.066179. Epub 2023 Oct 18. PMID 37850383